CLINICAL TRIAL: NCT01358461
Title: Circulating Biomarker(s) of Muscarinic Receptor Overexpression and Vagal Disorders.
Brief Title: Validation of a Non Invasive Blood Marker of SIDS and Vagal Disorders
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4900 (2010 - A01451-38)
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Vagal Syncope
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with vagal syncopes: Patients with vagal syncopes (n=120 : 60 adults & 60 children)
  Interventions: Biological: Blood sampling; Other: ECG-Holter 24 h tape and sino-carotid stimulation test
- Subjects controls without vagal syncopes: Subjects controls without vagal syncopes (n=120:60 adults & 60 children
  Interventions: Biological: Blood sampling; Other: ECG-Holter 24 h tape and sino-carotid stimulation test

INTERVENTIONS:
Biological: Blood sampling — Blood sampling
Other: ECG-Holter 24 h tape and sino-carotid stimulation test — ECG-Holter 24 h tape and sino-carotid stimulation test

SUMMARY:
Context

The investigators recently demonstrated a highly significant increase in muscarinic receptor density in the myocardium of infants deceased from sudden infant death syndrome (SIDS) compared to those of infants deceased from identified causes 1. Muscarinic receptor overexpression was found in all SIDS samples studied to date. It was associated with an average increase in acetylcholinesterase activity, appearing as a compensatory mechanism to oppose the cardiac muscarinic receptor overexpression. Similar vago-cardiac abnormalities were detected in a rabbit model of vagal hyperreactivity that the investigators first described some years ago2. In these hyperreactive animals, expression of muscarinic receptors was also enhanced in blood white cells. Noticeably, the pattern of changes in these cells paralleled the pattern of changes in the heart. Thus, muscarinic abnormalities in cardiac tissues could be inferred with high confidence from those measured in lymphocytes.This was the first report of a vago-cardiac abnormality in sudden infant death syndrome. The investigators findings also provided original and important perspectives for the identification and therapeutic management of infants at risk of sudden death. As such, the publication of the investigators work raised a major interest from the population and from the scientific and medical communities, in particular cardio-pediatricians. ObjectivesThe objective of the present clinical project is to validate, in human lymphocytes, muscarinic receptor expression level (assessed by quantitative RT-PCR) as a circulating biomarker of autonomic nervous system dysfunction and more specifically, of vagal hyperactivity and of risk of sudden death. The project will include 2 major items, conducted in parallel:1. evaluation of the muscarinic receptor expression in lymphocytes from adults with vagal syncopes (n=60 patients from an existing file versus 60 controls) (Cardiology unit + Clinical Investigation Centre (CIC) + Laboratory of Neurobiology and Cardiovascular Pharmacology); 2. evaluation of the muscarinic receptor expression in lymphocytes from children with vagal syncopes (n=60 versus 60 controls) (Pediatry unit + Clinical Investigation Centre + Laboratory of Neurobiology and Cardiovascular Pharmacology).PerspectivesThis project represents the first step of validation of a circulating marker of vagal hyperactivity and of risk of SIDS in human. Once this step is completed, the investigators will start with the prospective study " muscarinic receptor expression in lymphocytes and SIDS " (cord blood collected at birth and follow up of the new-borns) (Maternity ward + CIC + Laboratory of Neurobiology and Cardiovascular Pharmacology). Then therapeutic preventive management becomes a realistic objective. A therapeutic clinical study will then be started with atropinic drugs, in order to test their potential protective action against sudden death. The final objective of the investigators research is the prevention of SIDS through i) identification - as soon as birth - of new-borns at high risk and ii) appropriate prophylactic therapy. The investigators work also opens exciting perspectives in the field of the still poorly understood vagal disorders in children and adults such as vagal pauses.1 Livolsi et coll, Plos One 5, e9464, 2010 ; 2 Livolsi et coll, Circulation 106, 2301-2304, 2002

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 1 month to 50 years
* Patients with clinical signs of recurrent severe vagal syncopes
* Controls without clinical signs of recurrent severe vagal syncopes
* Mandatory clinical examination prior to enrolment

Exclusion Criteria:

* Autonomic nervous system disorders
* Cardiovascular, neurologic, psychiatric or metabolic diseases
* Drugs interfering with autonomic nervous system
* Doping or drug abuse
* Chronic smoking (more than 3 cigarettes a day
* Pregnancy

Ages: 1 Month to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo LIVOLSI, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France